CLINICAL TRIAL: NCT05919030
Title: Chemoradiation Versus Chemotherapy in Combination with Tislelizumab As First Line Treatment for Advanced Esophageal Squamous Cell Carcinoma with Low PD-L1 Expression (RENMIN-236): Multicentre, Randomised, Phase 3 Trial
Brief Title: A Study of Chemoradiation in Combination with Tislelizumab As First Line Treatment in Participants with Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yongshun Chen, Professor, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2023-K088
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Chemoradiation; Immunotherapy; Advanced esophageal cancer; Low PD-L1 expression; Progression-free survival
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy, Intensity-Modulated; tislelizumab; Cisplatin; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemoradiation + Tislelizumab (Experimental): Intensity-modulated radiotherapy (IMRT):
  Esophageal primary tumor: 39.6Gy/2.2Gy Bone metastasis: 30Gy/3Gy Lung, liver, brain metastases, metastatic lymph nodes: 45Gy/3Gy
  During concurrent radiation therapy:
  Drug: Tislelizumab 200 mg IV Q3W Drug: Nab Paclitaxel 75 mg/m² IV QW Drug: Cisplatin 25 mg/m² IV QW
  During consolidation therapy:
  Drug: Tislelizumab 200 mg IV Q3W Drug: Nab Paclitaxel 220 mg/m² IV Q3W Drug: Cisplatin 75 mg/m² IV Q3W
  Interventions: Radiation: Intensity-modulated radiotherapy (IMRT); Drug: Tislelizumab; Drug: Cisplatin; Drug: Nab paclitaxel
- Chemotherapy + Tislelizumab (Active Comparator): Drug: Tislelizumab 200 mg IV Q3W Drug: Nab Paclitaxel 220 mg/m² IV Q3W Drug: Cisplatin 75 mg/m² IV Q3W
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: Nab paclitaxel

INTERVENTIONS:
Radiation: Intensity-modulated radiotherapy (IMRT) — Esophageal primary tumor: 39.6Gy/2.2Gy Bone metastasis: 30Gy/3Gy Lung, liver, brain metastases, metastatic lymph nodes: 45Gy/3Gy
  Arms: Chemoradiation + Tislelizumab
Drug: Tislelizumab — 200 mg IV Q3W
Drug: Cisplatin — During concurrent radiation therapy: 25 mg/m² IV QW During consolidation therapy: 75 mg/m² IV Q3W
Drug: Nab paclitaxel — During concurrent radiation therapy: 75 mg/m² IV QW During consolidation therapy: 220 mg/m² IV Q3W

SUMMARY:
This study is a multicentre, randomised, parallel-controlled, open-label, 3 phase clinical trial. The subjects were untreated, unresectable locally advanced, recurrent or metastatic esophageal squamous cell carcinoma with low PD-L1 expression. Patients were randomly assigned to receive chemoradiation or chemotherapy in combination with Tislelizumab at a ratio of 1: 1. The primary endpoint was progression-free survival (PFS) in the intention-to-treat population. We hypothesized that in advanced esophageal squamous cell carcinoma patients with low PD-L1 expression, chemoradiation versus chemotherapy in combination with Tislelizumab will significantly improve PFS.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically confirmed squamous cell carcinoma of esophagus (per AJCC 8th edition).
2. Subjects must have unresectable advanced, recurrent or metastatic ESCC.
3. Subjects must not be amenable to curative approaches such as definitive chemoradiation and/or surgery.
4. PD-L1 expression (CPS) is less than 10.
5. No prior systemic anticancer therapy given as primary therapy for advanced or metastatic disease.
6. ECOG Performance Status of 0 or 1.
7. Subjects must have at least one measurable lesion by CT or MRI per RECIST 1.1 criteria; radiographic tumor assessment must be performed within 28 days prior to randomization.
8. Subjects must have adequate organ and bone marrow function.

Exclusion Criteria:

1. Presence of tumor cells in the brain or spinal cord which are symptomatic or require treatment.
2. Active known or suspected autoimmune disease.
3. Any serious or uncontrolled medical disorder or active infection.
4. Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
5. Any positive test result for hepatitis B or C indicating acute or chronic infection and/or detectable virus.
6. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Approximately 40 months from date of the first participant randomization
  PFS is defined as the time from the date of randomization to the date of first documentation of disease progression assessed by the investigator per RECIST v1.1 or death, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 40 months from date of the first participant randomization
  Overall Survival (OS) is defined as the time between the date of randomization and the date of death. For participants without documentation of death, OS will be censored on the last date the subject was known to be alive.
Objective Response Rate (ORR) | Approximately 40 months from date of the first participant randomization
  Objective response rate (ORR) is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). Best overall response (BOR) is defined as the best response designation as determined by BICR, recorded between the date of randomization and the date of objectively documented progression (per RECIST 1.1) or the date of subsequent anti-cancer therapy (including tumor-directed radiotherapy and tumor-directed surgery), whichever occurs first. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions. Complete response is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm.
Duration of Response (DOR) | Approximately 40 months from date of the first participant randomization
  DOR is defined as the time from the first determination of an objective response until the first documentation of progression assessed by the investigator per RECIST v1.1 or death, whichever comes first
Number of participants experiencing Adverse Events (AEs) | Approximately 40 months from date of the first participant randomization
  AEs are documented according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin hosptial of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No